CLINICAL TRIAL: NCT04333693
Title: Outcomes of Vascular Surgery in COVID-19 Infection: National Cohort Study (Covid-VAS)
Brief Title: Outcomes of Vascular Surgery in COVID-19 Infection: National Cohort Study
Acronym: Covid-VAS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Vascular Investigation Network Spanish Society for Angiology and Vascular Surgery (Network)
Responsible Party: Sponsor
Other Study IDs: RIV-2020-1
Record Dates: First submitted 2020-03-31; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Vascular Surgical Procedures; COVID-19; Postoperative Complications
Keywords: Vascular surgical procedures; Endovascular procedures; COVID-19; Postoperative complications; Prognosis
MeSH Terms: conditions — COVID-19; Postoperative Complications | interventions — Vascular Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Adults (age>18years) undergoing any type of vascular surgery (open surgery, endovascular surgery or hybrid procedure) in an operating theatre and either before or after surgery: lab test confirmed COVID-19 or clinical diagnosis of COVI-19 infection (no test performed)
  Interventions: Procedure: Vascular surgery

INTERVENTIONS:
Procedure: Vascular surgery — Open vascular, endovascular or hybrid procedures

SUMMARY:
There is an urgent need to understand the outcomes of COVID-19 infected patients who undergo surgery, specially vascular surgery. Capturing real-world data and sharing Spanish national experience will inform the management of this complex group of patients who undergo surgery throughout the COVID-19 pandemic, improving their clinical care.

The global community has recognised that rapid dissemination and completion of studies in COVID-19 infected patients is a high priority, so we encourage all stakeholders (local investigators, ethics committees, IRBs) to work as quickly as possible to approve this project.

This investigator-led, non-commercial, non-interventional study is extremely low risk, or even zero risk. This study does not collect any patient identifiable information (including no dates) and data will not be analysed at hospital-level.

DETAILED DESCRIPTION:
To determine 30-day mortality in patients with COVID-19 infection who undergo vascular surgery.

This will inform future risk stratification, decision making, and patient consent.

Inclusion criteria

The inclusion criteria are:

• Adults (age ≥18 years) undergoing ANY type of vascular surgery in an operating theatre, this includes open surgery, endovascular surgery or hybrid procedures.

AND

• Either before or after surgery: (i) lab test confirmed COVID-19 infection or (ii) clinical diagnosis of COVID-19 infection (no test performed).

Therefore this study should capture:

* emergency surgery patients with clinical diagnosis or lab confirmation of COVID-19 infection before surgery.
* emergency surgery patients with clinical diagnosis or lab confirmation of COVID-19 infection after surgery.
* elective surgery patients with clinical diagnosis or lab confirmation of COVID-19 infection after surgery. Patients who meet the inclusion criteria should be included regardless of surgical indication (aneurysm, limb or visceral ischemia, carotid stenosis, vascular trauma), anaesthetic type (local, regional, general), procedure type, or surgical approach (open surgery, endovascular surgery, hybrid procedure).

At most sites it is anticipated that the number of eligible patients is likely to be low. If possible all consecutive patients fulfilling inclusion criteria should be entered.

Study period Overall we plan to close data entry in September 2020 when the global pandemic is likely to be over, however individual centres may select their own study windows, depending on the timing of COVID-19 epidemic in their community.

Patient enrolment Ideally patients should be identified prospectively. However, given the rapid progression of the global pandemic, there may be no further new cases of COVID-19 infection in some hospitals that treated large numbers of COVID-19 earlier in the pandemic. It is important to capture the experience of these centres, therefore retrospective patient identification and data entry is permitted.

Primary outcome

* 30-day mortality Secondary outcome
* 7-day mortality
* 30-day reoperation
* Postoperative ICU admission
* Postoperative respiratory failure
* Postoperative acute respiratory distress syndrome (ARDS)
* Postoperative sepsis

Data collection Data will be collected and stored online through a secure server running the Spanish Society for Angiology and Vascular Surgery (SEACV) web application. This secure server allows collaborators to enter and store data in a secure system. A designated collaborator at each participating site will be provided with a project server login details, allowing them to securely submit data on to the system. Only anonymised data will be uploaded to the database. No patient identifiable data will be collected. Data collected will be on comorbidities, physiological state, treatment/operation, and outcome. No dates (e.g. date of surgery) will be collected. qSOFA and CURB-65 will be calculated based on the individual data points entered.

Local approvals The principal investigator at each participating site is responsible for obtaining necessary local approvals (e.g. research ethics committee or institutional review board approvals).The first approval will be on the Valladolid East Ethics Committee for Clinical Investigation.

Collaborators will be required to confirm that a local approval is in place at the time of uploading each patient record to the study database.

Where an audit approval is needed, this can be either registered as service evaluation, or to benchmark against an auditable standard (e.g. overall mortality after emergency surgery should be <15%).

Prior to formal local study approval, collaborators may prospectively collect data, but this should not be uploaded to the database until approval is confirmed.

Analysis A detailed statistical analysis plan will be written. Analyses will be overseen by the independent data monitoring committee (DMC). Reports will include description of the primary and secondary outcomes in the cohort. Multivariable modelling will be undertaken to CovidVAS protocol identify risk factors for 30-days mortality. Analyses will be stratified according to whether or not diagnosis of COVID-19 was confirmed by a lab test. Interim analyses will be performed as guided by the independent DMC. The first analysis will be performed once 50 patients have been entered on to the database, and the frequency of subsequent analyses will be agreed with the DMC. The decision to submit data for publication will be agreed by the steering committee with the DMC. Hospital-level data will not be released or published.

Authorship Collaborators from each site who contribute patients will be recognised on any resulting publications as PubMed-citable co-authors.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years) undergoing ANY type of vascular surgery in an operating theatre, this includes obstetrics. AND
* Either before or after surgery: (i) lab test confirmed COVID-19 infection or (ii) clinical diagnosis of COVID-19 infection (no test performed).

Therefore this study should capture:

* emergency surgery patients with clinical diagnosis or lab confirmation of COVID-19 infection before surgery.
* emergency surgery patients with clinical diagnosis or lab confirmation of COVID-19 infection after surgery.
* elective surgery patients with clinical diagnosis or lab confirmation of COVID-19 infection after surgery.

Exclusion Criteria:

* Not informed consent signed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COVID-19 infection who undergo vascular surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
30-days mortality | 30-days
  30-days mortality after vascular surgery in patients with COVID-19 infection

SECONDARY OUTCOMES:
7-days mortality | 7-days
  7-days mortality after vascular surgery in patients with COVID-19 infection
30-days reoperation | 30-days
  30-days reoperation after vascular surgery in patients with COVID-19 infection
Postoperative ICU admission | 30-days
  Postoperative ICU admission after vascular surgery in patients with COVID-19 infection
Postoperative respiratory failure | 30-days
  Postoperative respiratory failure after vascular surgery in patients with COVID-19 infection
Postoperative acute respiratory distress syndrome (ARDS) | 30-days
  Postoperative acute respiratory distress syndrome (ARDS) after vascular surgery in patients with COVID-19 infection
Postoperative sepsis | 30-days
  Postoperative sepsis after vascular surgery in patients with COVID-19 infection

CONTACTS AND LOCATIONS:
Locations (1):
- Spanish Society for Angiology and Vascular Surgery, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
No sharing plan available nowadays.

REFERENCES:
- [Background] Zoia C, Bongetta D, Veiceschi P, Cenzato M, Di Meco F, Locatelli D, Boeris D, Fontanella MM. Neurosurgery during the COVID-19 pandemic: update from Lombardy, northern Italy. Acta Neurochir (Wien). 2020 Jun;162(6):1221-1222. doi: 10.1007/s00701-020-04305-w. Epub 2020 Mar 28. No abstract available. PMID 32222820
- [Background] Aminian A, Safari S, Razeghian-Jahromi A, Ghorbani M, Delaney CP. COVID-19 Outbreak and Surgical Practice: Unexpected Fatality in Perioperative Period. Ann Surg. 2020 Jul;272(1):e27-e29. doi: 10.1097/SLA.0000000000003925. PMID 32221117
- [Background] Ficarra V, Novara G, Abrate A, Bartoletti R, Crestani A, De Nunzio C, Giannarini G, Gregori A, Liguori G, Mirone V, Pavan N, Scarpa RM, Simonato A, Trombetta C, Tubaro A, Porpiglia F; Research Urology Network (RUN). Urology practice during the COVID-19 pandemic. Minerva Urol Nefrol. 2020 Jun;72(3):369-375. doi: 10.23736/S0393-2249.20.03846-1. Epub 2020 Mar 23. PMID 32202401
- [Background] Iacobucci G. Covid-19: all non-urgent elective surgery is suspended for at least three months in England. BMJ. 2020 Mar 18;368:m1106. doi: 10.1136/bmj.m1106. No abstract available. PMID 32188602
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Derived] San Norberto EM, De Haro J, Pena R, Riera L, Fernandez-Caballero D, Sesma A, Rodriguez-Cabeza P, Ballesteros M, Gomez-Jabalera E, Taneva GT, Aparicio C, Moradillo N, Soguero I, Badrenas AM, Lara R, Torres A, Sala VA, Vaquero C; COVID-VAS Investigators from the Vascular Investigation Network (RIV) of the Spanish Society of Angiology and Vascular Surgery (SEACV). Outcomes After Vascular Surgery Procedures in Patients with COVID-19 Infection: A National Multicenter Cohort Study (COVID-VAS). Ann Vasc Surg. 2021 May;73:86-96. doi: 10.1016/j.avsg.2021.01.054. Epub 2021 Jan 22. PMID 33493590
- See also: Spanish Society for Angiology and Vascular Surgery — http://www.seacv.es